CLINICAL TRIAL: NCT03465826
Title: Developing a Mobile Health Pain-Coping Skills Training Program for the Treatment of Chronic Migraine: Testing Feasibility, Acceptability, and Utility, AIM 4
Brief Title: Developing a Mobile Health Pain-Coping Skills Training Program for the Treatment of Chronic Migraine: AIM 4
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Duke University (Other); Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 18-01218
Record Dates: First submitted 2018-02-02; First posted 2018-03-14 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Chronic Migraine, Headache
MeSH Terms: conditions — Headache | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PainCOACH Pain Coping Skills Training (Experimental): Migraineurs will participate in 4 weeks of daily headache monitoring, baseline questionnaires, followed by 8 weeks of the PainCOACH migraine mHealth Pain Coping Skills Training program (developed by Drs. Keefe and Rini based on social cognitive theory and in-person pain coping therapy sessions). Following the 8 week mHealth intervention, participants will immediately complete post-treatment assessments and later will complete follow-up assessments at 3 and 6 months.
  Interventions: Behavioral: PainCOACH Pain Coping Skills Training
- Treatment as Usual (Active Comparator): Participants will keep headache diaries for 4 weeks, followed by baseline assessments + 8 weeks of daily headache monitoring (as a parallel to the PainCOACH intervention). Post-assessments will immediately follow, and participants later will complete follow-up assessments at 3 and 6 months.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: PainCOACH Pain Coping Skills Training — Migraineurs will participate in 4 weeks of daily headache monitoring, baseline questionnaires, followed by 8 weeks of the PainCOACH migraine mHealth Pain Coping Skills Training program (developed by Drs. Keefe and Rini based on social cognitive theory and in-person pain coping therapy sessions). Following the 8 week mHealth intervention, participants will immediately complete post-treatment assessments and later will complete follow-up assessments at 3 and 6 months.
  Arms: PainCOACH Pain Coping Skills Training
Behavioral: Treatment as Usual — Participants will keep headache diaries for 4 weeks, followed by baseline assessments + 8 weeks of daily headache monitoring (as a parallel to the PainCOACH intervention). Post-assessments will immediately follow, and participants later will complete follow-up assessments at 3 and 6 months.
  Arms: Treatment as Usual

SUMMARY:
This ClinicalTrials.gov record pertains only to the clinical trial described below in Aim 4. Aims 1-3 and 5 are described here as background information. This study will be a two-site collaborative research effort (Wake Forest & Duke Univ.) drawing on expertise of investigators steeped in PCST, Internet-based treatment delivery, and development of cost-efficient and maximally-accessible behavioral interventions for migraine and chronic pain. This research will address four specific aims via a mixed-methods approach. In Aim 1 subjects (n=20) will be recruited to participate in user testing of the extant program (PainCOACH1). In Aim 2 subjects (n=64, including migraineurs, members of migraine patient advocacy groups, and clinical professionals trained in headache medicine) will participate in focus groups to provide guidance for appropriately tailoring the program for the treatment of chronic migraine. In Aim 3 feedback from Aims 1 and 2 will be employed to build and develop PainCOACH Migraine which will be beta-tested and refined. In Aim 4 subjects (n=144) will be recruited to participate in a randomized, controlled trial of the PainCOACH Migraine program (versus Medical Treatment as Usual) to demonstrate its feasibility, acceptability and engagement, and promise. Guided by findings from these aims a final exploratory aim will be conducted to optimize the program using prediction models to identify patients at risk for poor outcomes or attrition, and an adaptive therapeutic process targeting improved outcomes for such patients. Ultimately these research efforts will provide data and experience needed to support a subsequent large-scale and methodologically rigorous adaptive trial to test PainCOACH Migraine and enhance understanding of the potentials for Internet-based delivery of behavioral programs for individuals with chronic migraine.

DETAILED DESCRIPTION:
In addition to experiencing chronic pain, disability, and diminished quality of life, individuals with chronic migraine face critical access barriers to traditional, validated, clinic-based behavioral headache treatments (eg, availability of trained therapists, cost, absences from work). Internet-based and mHealth technologies show promise for the treatment of chronic pain conditions and are primed to address barriers to treatment, but have not yet been optimally translated into interventions for chronic migraine. A program of development is proposed to transform a validated, 8-week Internet-based pain-coping skills training (PCST) program (PainCOACH I; original) into a version specific for chronic migraine.

PainCOACH I was designed to retain key therapeutic components of in-clinic protocols and includes 8 modules of self-directed, tailored, interactive training in cognitive behavioral pain coping skills. A "virtual coach" provides verbal and visual instruction, feedback, and encouragement guided by theoretically-based learning principles. PainCOACH I has been successfully tested for populations with osteoarthritis and cancer pain, and has been studied in the US and Australia.

This clinical trial registration pertains only to Aim 4 of the study. In Aim 4 subjects (n=144) will be recruited to participate in a randomized, controlled trial of the PainCOACH Migraine program (versus Medical Treatment as Usual) to demonstrate its feasibility, acceptability and engagement, and promise.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Chronic migraine (diagnosed as 15 or more headaches per month)
* Willing and able to provide consent
* Able to speak and read English

Exclusion Criteria:

* headache disorder other than migraine
* change in preventive medications within 3 weeks prior to enrollment
* pain disorder other than migraine as a primary problem
* pregnant or planning pregnancy
* medical or psychiatric comorbidities likely to interfere with participation
* less than 7th grade reading proficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility and Engagement | Through study completion, an average of 9 months
  "Feasibility and Engagement" represent a single outcome measure that is measured using the PainCOACH Feasibility Questionnaire, which was developed by Co-Investigators Dr. Rini and Dr. Keefe for evaluating patients'experiences and satisfaction with PainCOACH. This measure has been used extensively in past and present studies conducted by their research teams and others. These instruments will be administered ONLY during the post-treatment assessment interval and includes both qualitative and quantitative survey items. Quantitative survey items will be scaled from 1 to 5 to indicate level of agreement, where "1" indicates "strong agreement" and "5" indicates "strong disagreement".

SECONDARY OUTCOMES:
Change in Migraine Disability | Baseline, 2 months, 5 months, and 8 months
  The MIDAS (NINDS CDE 2.0 "highly recommended") was developed to assess headache-related disabilities focusing on care for persons with migraine [[Stewart 2000, 2001]]. Headache sufferers answer 5 questions (self-administered) related to the last 3 months, indicating the number of days their everyday life has been limited by migraines. MIDAS assesses disability in 3 areas: a) household work, b) paid work and/or school, and c) social, leisure, and family activities. MIDAS is valuable for quantification of headache disability and as a reference for measuring improvement. The MIDAS is widely employed, internally consistent, highly reliable, valid, and correlates with physicians' clinical judgments. The instrument usually takes less than 5 minutes to complete and is easy to understand.
Change in HIT-6 | Baseline, 2 months, 5 months, and 8 months
  The HIT-6 (NINDS CDE 2.0 "highly recommended") is a 6-question self-report tool that measures the impact headaches have on a person's ability to function on the job, at home, at school, and in social situations, with items that address a spectrum of health outcomes (ranging from pain to emotional distress)81,82. The HIT-6 is widely use and well validated, and employs a recall period of 4 weeks
Change in pain intensity | Baseline, 2 months, 5 months, and 8 months
  The Pain NRS (Numeric Rating Scale) will be used to assess pain intensity and to facilitate comparison of findings across trials examining PainCOACH. Specifically, patients are asked to rate average, worst, and least levels of pain intensity over the past week on a scale with ratings ranging from 0 "no pain" to 10 "worst possible pain." Minimally, moderately, and substantially important clinical change are represented by a decrease in score by 10% to 20%, >=30%, and >=50%, respectively80. The Pain NRS has been validated as a treatment outcome measure and is recommended as a core outcome measure of clinical trials in chronic pain patients at the IMPAACT-II consensus meeting.
Change in headache management self-efficacy | Baseline, 2 months, 5 months, and 8 months
  The HMSE (Headache Management Self-Efficacy scale) is a 25-item headache-specific measure of self-efficacy employing Likert-type rating scale ranging from 1 to 7 with questions in order to quantify headache patients' confidence in their own ability to prevent and manage headache attacks. The HMSE is established as both reliable and valid.
Change in headache locus of control scale | Baseline, 2 months, 5 months, and 8 months
  The HSLC (Headache-Specific Locus of Control Scale) is a 33-item self-report questionnaire designed specifically for recurrent headache sufferers to assess the individual's perceptions that headache problems and headache relief are determined primarily by the individual's behavior (Internal Locus of Control), the actions of health care professionals (Health Care Professionals Locus of Control), or chance factors (Chance Locus of Control). The Likert-type item responses range from 1 (strongly disagree) to 5 (strongly agree). Factor analysis confirmed the 3-factor structure of the HSLC, and the reliability of the subscales is established (Cronbach ́s α of .86, .84 and .88 for each factor, respectively) and confirmed.
Change in pain catastrophizing | Baseline, 2 months, 5 months, and 8 months
  The PCS (Pain Catastrophizing Scale) is a 13-item self-report measure of the tendency to ruminate, magnify, or feel hopeless about, that is, catastrophize about pain. Each item is rated on a 5-point scale ranging from 0 "not at all" to 4 "all the time," with a total summed scale score ranging from 0 to 52. A score of >=30 is suggestive of clinically relevant levels of catastrophizing. The PCS was administered at the beginning of each session.

CONTACTS AND LOCATIONS:
Overall Officials: Donald B Penzien, PhD, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No